CLINICAL TRIAL: NCT00518323
Title: A Randomized, Multicenter, Double-Blind, Weight-Based, Fixed-Dose, Parallel-Group, Placebo-Controlled Study of the Efficacy and Safety of Extended Release Paliperidone for the Treatment of Schizophrenia in Adolescent Subjects, 12 to 17 Years of Age
Brief Title: A Double-blind, Placebo-controlled Study of the Safety and Efficacy of Paliperidone Extended Release (ER) in the Treatment of Schizophrenia in Adolescent Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR002368; R076477PSZ3001
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 001 (Experimental): Paliperidone ER 1.5 mg tablet once daily for 6 weeks
  Interventions: Drug: Paliperidone ER
- 002 (Experimental): Paliperidone ER 3 mg or 6 mg tablet once daily for 6 weeks
  Interventions: Drug: Paliperidone ER
- 003 (Experimental): Paliperidone ER 6 mg or 12 mg tablet once daily for 6 weeks
  Interventions: Drug: Paliperidone ER
- 004 (Placebo Comparator): Placebo Once daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paliperidone ER — 3 mg or 6 mg tablet once daily for 6 weeks
  Arms: 002
Drug: Placebo — Once daily for 6 weeks
  Arms: 004
Drug: Paliperidone ER — 1.5 mg tablet once daily for 6 weeks
  Arms: 001
Drug: Paliperidone ER — 6 mg or 12 mg tablet once daily for 6 weeks
  Arms: 003

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of 3 weight-based, fixed-dose groups of paliperidone extended release (ER) compared with placebo in adolescent patients between 12 to 17 years of age, who are diagnosed with schizophrenia. Paliperidone ER is an atypical antipsychotic agent approved by the U.S. Food and Drug Administration for the treatment of schizophrenia in adults. Patients may be voluntary inpatients or outpatients at the time of the screening visit, but should have returned to their usual living situation by Day 21 of the double-blind treatment phase. The study duration is approximately 10 weeks. Patients who have completed this study or who were discontinued from this study due to lack of efficacy but have completed at least 21 days of double-blind treatment and are expected to benefit from paliperidone treatment, may enter an optional open-label safety study.

DETAILED DESCRIPTION:
The study is a multicenter, randomized (treatment group is assigned by chance), double-blind (neither the physician nor the patient knows which treatment group the patient is in), parallel-group, placebo controlled study. This study will enroll adolescent men and women who have schizophrenia as specified by the Diagnostic and Statistical Manual of Mental Disorders; 4th Edition (DSM-IV) diagnosis of schizophrenia (295.10, 295.20, 295.30, 295.60, and 295.90) as confirmed by the Kiddie-Sads-Present and Lifetime Version (KSADS-PL), and who should have a Positive and Negative Syndrome Scale (PANSS) score that is between 60 and 120, inclusive, at screening and baseline. Before any study related procedure is performed, the patient and his parent or legal guardian must have provided assent and signed an informed consent form, respectively. The study consists of 3 phases: a screening phase, a 6-week double-blind treatment phase with an end-of-study or early withdrawal visit, and a 1 week follow-up visit for patients who do not enter the optional open-label safety study. In the screening phase, a trained clinician will complete the K SADS-PL interview, including all 5 supplements, to confirm the DSM-IV diagnostic criteria for schizophrenia. In addition, the K-SADS-PL screening diagnostic interview items for suicide must each have a score of <=2, as follows: item a), recurrent thoughts of death; item b), suicidal thoughts; item c), suicide attempts and their seriousness; item d), suicide attempts and their lethality; and item e) self harming behavior. Women of childbearing potential will undergo a urine pregnancy test at screening, baseline, Week 4, and at end of study or upon early withdrawal from the study. Patients who are receiving prohibited medications, such as antidepressants, lithium, drugs of abuse, and alcohol, will enter a washout period during which medications will be tapered down and eventually stopped. The screening and washout phase may not exceed 21 days. In the double-blind treatment phase, at the baseline visit, the inclusion and exclusion criteria will be reviewed. Patients who continue to meet the criteria will be randomly assigned (as in the toss of a coin) to 1 of 4 dose groups. Patients weighing between 29 to <51 kilograms (kg) will receive paliperidone ER 1.5, 3.0, or 6.0 milligrams (mg) or matching placebo. Patients weighing >=51 kg will receive paliperidone ER 1.5, 6.0, or 12.0 mg or matching placebo. Patients will come to the study site for weekly visits during this phase. A follow-up visit will occur 1 week after the end of treatment for those patients who will not enter the open-label study. Efficacy and safety procedures will be performed at specified times during the study. Efficacy procedures include the administration of the PANSS, Children's Global Assessment (CGAS), Clinical Global Impression-Severity (CGI-S) and a sleep visual analog scale. Safety assessments include a physical examination (ECG measurements, vital signs, weight, height, and waist measurements), clinical laboratory testing, drug screen, Simpson and Angus Scale (SAS), Barnes Akathisia Rating Scale (BARS), Abnormal Involuntary Movement Scale (AIMS), Tanner Staging, concomitant medications and the recording of adverse events. A Data Safety Monitoring Board will oversee the conduct of the study and review adverse event reports and laboratory test results. The total volume of blood drawn for laboratory evaluation throughout the study, including 10 milliliters (mL) for the optional pharmacogenomics testing, is approximately 66 mL for each patient. Blood samples will be collected to explore the pharmacokinetics of paliperidone in adolescent patients. The study hypothesis is that at least 1 paliperidone ER dose group will be superior to placebo in improving the symptoms of schizophrenia as measured by the change in total PANSS score from the baseline to endpoint (Week 6). Paliperidone ER 1.5, 3.0, 6.0, or 12.0 mg or matching placebo will be administered daily in the morning before 10 a.m., and at approximately the same time each day. Study drug administration should occur in a consistent manner relative to the intake of food (i.e., either before or after breakfast, or without any breakfast) throughout the study. Study drug should be swallowed whole and with water. Study drug will be administered for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV) criteria for schizophrenia (295.10, 295.20, 295.30, 295.60, 295.90) for 1 year (the diagnosis will be established using the K-SADS-PL, including all supplements)
* Must not be a danger to themselves or others, and must have family support available to be maintained as an outpatient
* Should have had at least 1 adequate treatment with an antipsychotic before participation in this study
* Must have a PANSS score between 60 and 120, inclusive, at screening and baseline
* Weight >=29 kg

Exclusion Criteria:

* Meet the DSM-IV criteria at screening for dissociative disorder, bipolar disorder, major depressive disorder, schizoaffective disorder, schizophreniform disorder, autistic disorder, or primary substance induced psychotic disorder. Other comorbid disorders e.g., attention-deficit hyperactivity disorder (ADHD) are allowed as long as the diagnosis of schizophrenia is the primary diagnosis and the comorbid disorders in the investigator's judgment do not require medication
* Mild, moderate, or severe mental retardation (i.e., documented intelligence quotient [IQ] <70) established by previous IQ testing or history
* Women who are pregnant (as confirmed by urine pregnancy test performed at screening or baseline), planning to become pregnant or are nursing
* Have a known or suspected history of seizure disorder, or neuroleptic malignant syndrome, encephalopathic syndrome, tardive dyskinesia, or insulin dependent diabetes mellitus
* Presence of any significant or unstable cardiovascular, respiratory, renal, hepatic, hematologic, endocrine, immunologic, or other systemic disease

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (34):
- United States (10):
  - Cerritos, California
  - Fountain Valley, California
  - San Diego, California
  - Santa Ana, California
  - Washington D.C., District of Columbia
  - Lake Charles, Louisiana
  - Boston, Massachusetts
  - Cleveland, Ohio
  - Portsmouth, Virginia
  - Spokane, Washington
- India (7):
  - Bangalore
  - Chennai
  - Hyderabad
  - Hyderabad Andra Pradesh
  - Mangalore
  - New Delhi
  - Varanasi
- Bucharest, Romania
- Russia (11):
  - Ekaterinburg Na
  - Kazan'
  - Moscow
  - Moscow Russia
  - Nizhny Novgorod
  - Saint Petersburg
  - Saratov
  - Smolensk Region N/A
  - Stavropol Na
  - Tomsk Na
  - Yaroslavl
- Ukraine (5):
  - Hlevakha
  - Kharkiv
  - Kiev
  - Odesa
  - Simferopol

REFERENCES:
- [Derived] Sliwa JK, Fu DJ, Bossie CA, Turkoz I, Alphs L. Body mass index and metabolic parameters in patients with schizophrenia during long-term treatment with paliperidone palmitate. BMC Psychiatry. 2014 Feb 22;14:52. doi: 10.1186/1471-244X-14-52. PMID 24559194
- [Derived] Opler M, Malaspina D, Gopal S, Nuamah I, Savitz AJ, Singh J, Hough D. Effect of parental age on treatment response in adolescents with schizophrenia. Schizophr Res. 2013 Dec;151(1-3):185-90. doi: 10.1016/j.schres.2013.10.001. Epub 2013 Oct 18. PMID 24144440
- See also: A double-blind, placebo-controlled study of the safety and efficacy of paliperidone extended release (ER) in the treatment of schizophrenia in adolescent patients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=55&filename=CR002368_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started 8 August 2007 in medical clinics located around the world. The study ended on 30 March 2009.
Pre-assignment Details: Subjects who were eligible for the study had their current disallowed psychotropic medications washed out prior to assignment to treatment groups. Subjects who violated inclusion criteria before assignment (eg, because they continued to take a disallowed medication) were to be removed from the study.
Groups:
- Pali ER Low: Paliperidone ER 1.5 mg for subjects weighing 29 kg and above
- Pali ER Medium: Paliperidone ER 3 mg (for subjects weighing between 29 kg and less than 51 kg) or 6 mg (for subjects weighing 51 kg and above)
- Pali ER High: Paliperidone ER 6 mg (for subjects weighing between 29 kg and less than 51 kg) or 12 mg (for subjects weighing 51 kg and above)
Period: Overall Study
Arm/Group | Pali ER Low | Pali ER Medium | Pali ER High | Placebo
Started | 54 | 48 | 48 | 51
Completed | 35 | 40 | 37 | 26
Not Completed | 19 | 8 | 11 | 25
Not completed — Lack of Efficacy | 14 | 2 | 4 | 20
Not completed — Withdrawal by Subject | 1 | 2 | 4 | 2
Not completed — Lost to Follow-up | 0 | 2 | 1 | 3
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Prohibited medication and others | 3 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pali ER Low | Pali ER Medium | Pali ER High | Placebo | Total
Number analyzed (Participants) | 54 | 48 | 48 | 51 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54 | 48 | 48 | 51 | 201
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.50) | 15.3 (1.60) | 15.5 (1.60) | 15.7 (1.40) | 15.4 (1.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 17 | 14 | 28 | 83
  Male | 30 | 31 | 34 | 23 | 118
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 7 | 9 | 30
  Ukraine | 9 | 8 | 9 | 8 | 34
  Romania | 2 | 3 | 3 | 2 | 10
  Russian Federation | 22 | 20 | 19 | 21 | 82
  India | 13 | 11 | 10 | 11 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in the PANSS Total Score From Baseline to the Last Postrandomization Assessment in the Double-blind Period of the Study.
Description: The Positive and Negative Syndrome Scale (PANSS) measures the severity of psychotic symptoms of schizophrenia. Scores range from 30 to 210, where 30=best and 210=worst. The change in PANSS total score for all eligible subjects was measured from the beginning of the study to the end.
Time Frame: 6 weeks
Population: The number of participants in the intent-to-treat (ITT) analysis set was used. This set includes patients who received study drug and have at least 1 efficacy measurement. The Last Observation Carried Forward method was used for imputation; ie, the last measure for subjects who ended study early was carried forward as if they completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pali ER Low | Pali ER Medium | Pali ER High | Placebo
Number analyzed (Participants) | 54 | 48 | 47 | 51
units on a scale | -9.8 (16.31) | -17.3 (14.33) | -13.8 (15.74) | -7.9 (20.15)
Statistical Analysis 1: Comparison: Pali ER Low vs Placebo; If there were approximately 49 subjects per treatment group who had Week 6 (LOCF or end point) PANSS total measurements, the study was expected to have approximately 80% power to detect a clinically relevant difference of 13.2 points between any paliperidone ER group compared with placebo for the primary outcome measure; Test type: Superiority or Other; p = 0.508, ANCOVA — The p value was associated with the closed testing procedure using Dunnett's test; Used ANCOVA model with treatment(placebo, pali ER Low, pali ER Medium, and pali ER High) and country as factors and baseline value as a covariate; Mean Difference (Final Values) = -2.1, 95% CI [-8.36 to 4.16], Standard Error of Mean 3.17 — The 95% confidence intervals were unadjusted for multiplicity
Statistical Analysis 2: Comparison: Pali ER Medium vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.006, ANCOVA — The p value was associated with the closed testing procedure using Dunnett's test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.1, 95% CI [-16.58 to -3.67], Standard Error of Mean 3.27 — The 95% confidence intervals were unadjusted for multiplicity
Statistical Analysis 3: Comparison: Pali ER High vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.086, ANCOVA — The p value was associated with the closed testing procedure using Dunnett's test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.6, 95% CI [-13.07 to -0.09], Standard Error of Mean 3.29 — The 95% confidence intervals were unadjusted for multiplicity

2. Secondary Outcome: Change From Baseline to End Point in Clinical Global Impression-Severity (CGI-S) Scale
Description: The CGI-S rating scale was used to assess the severity of a subject's overall clinical condition. Scores range from 1 to 7, where 1=best and 7=worst.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pali ER Low | Pali ER Medium | Pali ER High | Placebo
Number analyzed (Participants) | 54 | 48 | 47 | 51
units on a scale | 0.0 [-3.00 to 1.00] | -1.0 [-3.00 to 0.00] | -1.0 [-3.00 to 1.00] | 0.0 [-3.00 to 1.00]
Statistical Analysis 1: Comparison: Pali ER Low vs Placebo; Analysis of the change in the CGI-S score at end point was performed using an analysis of covariance model on the ranks of the change in score at end point with treatment (placebo, pali ER Low, pali ER Medium, and pali ER High) and country as factors, and (non-ranked) baseline CGI-S score as a covariate; Test type: Superiority or Other; p = 0.968, ANCOVA — Comparison with placebo was without multiplicity adjustment
Statistical Analysis 2: Comparison: Pali ER Medium vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison with placebo was without multiplicity adjustment
Statistical Analysis 3: Comparison: Pali ER High vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.021, ANCOVA — Comparison with placebo was without multiplicity adjustment

3. Secondary Outcome: Change From Baseline to End Point in Children's Global Assessment (CGAS) Score
Description: The CGAS score assesses psychological, social, and school functioning for children 6 to 17 years of age. Scores range from 1 to 100, where 100=best and 1=worst.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pali ER Low | Pali ER Medium | Pali ER High | Placebo
Number analyzed (Participants) | 54 | 48 | 47 | 51
units on a scale | 4.4 (10.72) | 13.1 (12.07) | 8.6 (11.18) | 5.0 (13.82)
Statistical Analysis 1: Comparison: Pali ER Low vs Placebo; Test type: Superiority or Other; p = 0.846, ANCOVA — Comparison with placebo was without multiplicity adjustment; Used ANCOVA model with treatment (placebo, pali ER Low, pali ER Medium, and pali ER High) and country as factors and baseline value as a covariate; Mean Difference (Final Values) = -0.4, 95% CI [-4.54 to 3.73], Standard Error of Mean 2.10
Statistical Analysis 2: Comparison: Pali ER Medium vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison with placebo was without multiplicity adjustment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.6, 95% CI [4.28 to 12.82], Standard Error of Mean 2.17
Statistical Analysis 3: Comparison: Pali ER High vs Placebo; Test type: Superiority or Other; p = 0.067, ANCOVA — Comparison with placebo was without multiplicity adjustment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.0, 95% CI [-0.28 to 8.33], Standard Error of Mean 2.18

4. Secondary Outcome: Change From Baseline to End Point in Sleep Visual Analog Scale (VAS) for Quality of Sleep.
Description: The sleep VAS for sleep quality is a scale for measuring the quality of sleep experienced by a patient. Scores range from 0 to 100, where 100=best and 0=worst.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pali ER Low | Pali ER Medium | Pali ER High | Placebo
Number analyzed (Participants) | 54 | 48 | 47 | 50
units on a scale | 6.6 (24.57) | 16.0 (27.06) | 14.4 (22.72) | -0.3 (34.21)
Statistical Analysis 1: Comparison: Pali ER Low vs Placebo; Test type: Superiority or Other; p = 0.058, ANCOVA — Comparison with placebo was without multiplicity adjustment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.1, 95% CI [-0.29 to 16.56], Standard Error of Mean 4.27
Statistical Analysis 2: Comparison: Pali ER Medium vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison with placebo was without multiplicity adjustment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 16.8, 95% CI [8.08 to 25.43], Standard Error of Mean 4.40
Statistical Analysis 3: Comparison: Pali ER High vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — Comparison with placebo was without multiplicity adjustment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 13.5, 95% CI [4.76 to 22.23], Standard Error of Mean 4.43

5. Secondary Outcome: Change From Baseline to End Point in Sleep VAS for Daytime Drowsiness
Description: The sleep VAS for daytime drowsiness is a scale for measuring the drowsiness experienced by a patient. Scores range from 0 to 100, where 100=best and 0=worst.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pali ER Low | Pali ER Medium | Pali ER High | Placebo
Number analyzed (Participants) | 54 | 48 | 47 | 50
units on a scale | -6.2 (24.69) | -7.2 (25.22) | 1.0 (29.55) | -2.8 (30.27)
Statistical Analysis 1: Comparison: Pali ER Low vs Placebo; Test type: Superiority or Other; p = 0.237, ANCOVA — Comparison with placebo was without multiplicity adjustment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.9, 95% CI [-13.11 to 3.26], Standard Error of Mean 4.15
Statistical Analysis 2: Comparison: Pali ER Medium vs Placebo; Test type: Superiority or Other; p = 0.119, ANCOVA — Comparison with placebo was without multiplicity adjustment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.7, 95% CI [-15.15 to 1.74], Standard Error of Mean 4.28
Statistical Analysis 3: Comparison: Pali ER High vs Placebo; Test type: Superiority or Other; p = 0.574, ANCOVA — Comparison with placebo was without multiplicity adjustment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.4, 95% CI [-11.00 to 6.11], Standard Error of Mean 4.34

ADVERSE EVENTS:
Arm/Group | Pali ER Low | Pali ER Medium | Pali ER High | Placebo
Serious Adverse Events (participants affected / at risk) | 2/54 | 1/48 | 1/48 | 1/51
Other Adverse Events (participants affected / at risk) | 19/54 | 20/48 | 33/48 | 24/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pali ER Low (N=54) | Pali ER Medium (N=48) | Pali ER High (N=48) | Placebo (N=51)
Schizophrenia (Psychiatric disorders) | 1 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pali ER Low (N=54) | Pali ER Medium (N=48) | Pali ER High (N=48) | Placebo (N=51)
Somnolence (Nervous system disorders) | 3 | 7 | 10 | 1
Akathisia (Nervous system disorders) | 2 | 4 | 8 | 0
Headache (Nervous system disorders) | 5 | 3 | 5 | 2
Cogwheel rigidity (Nervous system disorders) | 0 | 0 | 4 | 0
Dystonia (Nervous system disorders) | 1 | 1 | 4 | 0
Tremor (Nervous system disorders) | 1 | 4 | 4 | 0
Insomnia (Psychiatric disorders) | 5 | 3 | 6 | 11
Anxiety (Psychiatric disorders) | 0 | 0 | 4 | 2
Schizophrenia (Psychiatric disorders) | 5 | 0 | 2 | 4
Agitation (Psychiatric disorders) | 3 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 4 | 6
Vomiting (Gastrointestinal disorders) | 0 | 3 | 4 | 5
Tachycardia (Cardiac disorders) | 0 | 2 | 4 | 0
Weight increased (Investigations) | 4 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3

LIMITATIONS AND CAVEATS:
No information about longer-term (ie, >6 weeks) efficacy and safety in adolescents or in young (<12 years) children with schizophrenia. Results with doses less than 1.5 mg or more than 12 mg cannot be extrapolated from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days